CLINICAL TRIAL: NCT03077295
Title: Role of Breakfast Size and Composition for Appetite Control and Energy Balance
Brief Title: The Big Breakfast Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aberdeen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 804
Record Dates: First submitted 2016-12-01; First posted 2017-03-10 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-06

CONDITIONS: Obesity; Weight Loss
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Fibre to High-Protein (HF-HP) (Experimental): * Phase 1: no intervention, habitual diet for 4 days and then 3day maintenance diet
  * Phase 2: consumption of HF meals for 4 weeks
  * Phase 3: washout for 1 week, controlled maintenance diet
  * Phase 4: consumption of HP meals for 4 weeks
  Interventions: Other: High Fibre; Other: High Protein
- High Protein to High-Fibre (HP-HF) (Experimental): * Phase 1: no intervention, habitual diet for 4 days and then 3day maintenance diet
  * Phase 2: consumption of HP meals for 4 weeks
  * Phase 3: washout for 1 week, controlled maintenance diet
  * Phase 4: consumption of HF meals for 4 weeks
  Interventions: Other: High Fibre; Other: High Protein

INTERVENTIONS:
Other: High Fibre — High fibre/carbohydrate (50% CHO, 35% fat and 15% Protein) with 45% calories at breakfast and 20% evening meal provided and buffet lunch. Total dietary fibre will be at least 30g/d for 2000kcal intake and provided as a mixed soluble and insoluble fibre sources to maintain palatability of the diet (e.g. wheat bran, fava bean, lentil, buckwheat).
  Other Names: HF
Other: High Protein — • High protein diet (30% protein, 35% fat and 35% CHO) with 45% calories at breakfast and 20% evening meal provided and buffet lunch. Protein will be a mixed meat matrix to include poultry, fish, red meat, prawns, eggs, dairy. Total dietary fibre will be no more than 15g/d for 2000kcal intake.
  Other Names: HP

SUMMARY:
This weight loss study will investigate the impact of diet composition and meal size (large breakfast meals and smaller evening meals) on body weight, energy balance and eating behaviour, by altering calorie (meal) distribution.

DETAILED DESCRIPTION:
The aim of this study is to further strengthen our understanding of the role of dietary components (in particular fibre and protein) in a healthy diet. The information gained from this research will lead to better policy advice, particularly in relation to healthy weight management, metabolic control, mental health and intestinal health. It will also lay the foundations to produce healthier primary products and aid the food industry in developing new and healthier products (e.g. products that aid hunger control and satiety). This will be addressed through four interlinked objectives:

O1: Healthy weight management and improved metabolic and mental health O2: Identification of gut bacteria and compounds of relevance to vascular and gut health O3: Linking fibre consumption to intestinal microbial communities and health O4: Mathematical modelling of interactions between diet and gut microbial communities

ELIGIBILITY:
Inclusion Criteria:

* BMI ranging from 27-42 kg/m2;
* those habitually consuming breakfast (at least 5 times a week).

Exclusion Criteria:

* women who are pregnant, planning to be pregnant or breastfeeding
* subjects with food allergy
* diagnosis of diabetes, hypertension, renal, hepatic, haematological disease or coronary heart disease
* having given a pint of blood for transfusion purposes within the last month
* unsuitable veins for blood sampling
* inability to understand the participant information sheet
* inability to speak, read and understand the English language
* those on any prescription medications (other than oral contraceptives)
* those on any specific diet regimes
* those on any weight loss programmes (that may be affecting lifestyle, physical activity and diet).

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2017-04-05 (Actual); Primary Completion 2019-04-05 (Actual); Study Completion 2019-04-05 (Actual)

PRIMARY OUTCOMES:
Change in Energy Balance | measured up to day 71 of study
  Chronic influence on energy balance (body weight, kg)

SECONDARY OUTCOMES:
Acute effects on appetite after test meals | Baseline & week 4 of each treatment
  Appetite questionnaires recorded on Visual Analogue Scales every 30mins on test days
Acute effects on biomarkers of health after test meals | Baseline & week 4 of each treatment
  blood samples analysed for Glucose, Lipids and Hormones
Acute effects on gastric emptying after test meals | Baseline & week 4 of each treatment
  gastric emptying (stable isotope, Octanoic acid labelled breath samples)
Resting Metabolic Rate (RMR) before & after test meals | Baseline & week 4 of each treatment
  Chronic influence on metabolism or Thermic Effect of Food (TEF) using indirect calorimetry measurement
Faecal sample analysis for gut health | up to 10 weeks
  Chronic influence on changes in gut microbiota
Bone Density | Baseline & week 4 of each treatment
  Dual Energy X-ray Absorptiometry (DXA) Scan to measure fat mass, fat free mass & bone density as part of the 4 compartment model
Body Composition | Baseline & week 4 of each treatment
  Air Displacement Plethysmography (BodPod) to measure body fat as part of the 4 compartment model
Total Body Water | Baseline & week 4 of each treatment
  Deuterium Dilution to measure Total Body Water (TBW) as part of the 4 compartment model

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Johnstone, PhD, Principal Investigator — Senior Research Fellow
Locations (1):
- The Rowett Institute, Aberdeen, United Kingdom

IPD SHARING:
Plan to Share IPD: No